CLINICAL TRIAL: NCT00658138
Title: Clinical Evaluation of 3M™ ESPE™ Adper™ Scotchbond™ SE Self-Etch Adhesive in Class I and Class II Restorations in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-07-020
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adhesive A (Experimental)
  Interventions: Device: 3M ESPE Adper Scotchbond SE
- Adhesive B (Active Comparator)
  Interventions: Device: 3M ESPE Adper Scotchbond 1XT

INTERVENTIONS:
Device: 3M ESPE Adper Scotchbond SE — To be used per manufacturer's instructions.
  Other Names: Dental adhesive used for bonding fillings
  Arms: Adhesive A
Device: 3M ESPE Adper Scotchbond 1XT — To be used per manufacturer's instructions.
  Other Names: Dental adhesive used for bonding fillings
  Arms: Adhesive B

SUMMARY:
The purpose of this study is to evaluate the performance of a new dental adhesive system in the restoration of Class I and Class II cavities in adult teeth.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age
* Must have 2 or 4 qualifying Class I or Class II cavities
* Must be willing to sign consent form
* Must be willing to return to University dental clinic for 4 study appointments
* Must be in good medical health and able to tolerate dental procedures

Exclusion Criteria:

* Current participation in other restorative product studies
* Known allergies to dental products
* Unacceptable level of oral hygiene
* Chronic periodontitis (gum disease)
* Rampant caries (cavities)
* Severe salivary gland problems
* Inability or unwillingness to attend study appointments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-12; Primary Completion 2010-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Dondi dall'Orologio, Professor, Principal Investigator — University of Bologna
Locations (1):
- University of Bologna, Clinica Odontoiatrica, Bologna, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 61 subjects were recruited from 70 patients with a total of 134 study teeth. Recruitment was from December 2008 to April 2009. Subjects were recruited from patients attending PI's clinic
Pre-assignment Details: All enrolled participants took part in the study
Groups:
- 3M ESPE Adper Scotchbond SE and 3M ESPE Adper Scotchbond 1XT: 67 teeth in 61 subjects had 3M ESPE Adper Scotchbond SE 67 teeth in 61 subjects had 3M ESPE Adper Scotchbond 1XT
Period: Overall Study
Arm/Group | 3M ESPE Adper Scotchbond SE and 3M ESPE Adper Scotchbond 1XT
Started | 61
Completed | 40
Not Completed | 21

BASELINE CHARACTERISTICS:
Arm/Group | 3M ESPE Adper Scotchbond SE and 3M ESPE Adper Scotchbond 1XT
Number analyzed (Participants) | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 61
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 27
Region of Enrollment [Number; unit: participants]
  Italy | 61

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Restorations Scoring Alpha
Description: Restorations were scored Alpha, Bravo or Charlie for retention, post-operative sensitivity, anatomic form, margin integrity, color match, stain resistance, and secondary caries. Alpha score = 'excellent' Bravo = 'acceptable' Charlie = 'unsatisfactory'. Total Alpha scores were evaluated for the primary outcome.
Time Frame: 12 months
Population: Analysis was based on the number of study teeth available for review at 12 months
Measure: Number; unit: percentage of Alpha scores
Units Other Than Participants: restorations
Groups:
- Scotchbond SE: 3M ESPE Adper Scotchbond SE
- Scotchbond 1XT: 3M ESPE Adper Scotchbond 1XT
Arm/Group | Scotchbond SE | Scotchbond 1XT
Number analyzed (Participants) | 40 | 40
Number analyzed (restorations) | 46 | 46
percentage of Alpha scores | 100 | 96
Statistical Analysis 1: Comparison: Scotchbond SE vs Scotchbond 1XT; Hypothesis was no difference between adhesives tested at one year. Restorations were scored using USPHS subjective clinical criteria; Test type: Non-Inferiority or Equivalence — No power calculation done - pilot study; p = 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.05
Statistical Analysis 2: Comparison: Scotchbond SE vs Scotchbond 1XT; Null hypothesis is adhesives are not different in clinical performance at one year; Test type: Non-Inferiority or Equivalence — No power calculation done - pilot study; p > 0.05, Wilcoxon (Mann-Whitney); percentage of Alpha values

ADVERSE EVENTS:
Time Frame: One year
Arm/Group | 3M ESPE Adper Scotchbond SE and 3M ESPE Adper Scotchbond 1XT
Serious Adverse Events (participants affected / at risk) | 0/61
Other Adverse Events (participants affected / at risk) | 0/61

LIMITATIONS AND CAVEATS:
Main limitation of study was small sample size and short duratrion. Study was a pilot of one year's duration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No